CLINICAL TRIAL: NCT06481098
Title: A Randomized, Double-Blind, Placebo-Controlled, Single- and Multiple-Ascending Dose Study to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of HM15275 in Healthy and Obese Subjects
Brief Title: A Phase 1 Study to Assess HM15275 in Healthy and Obese Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: HM-OBCT-101
Record Dates: First submitted 2024-05-30; First posted 2024-07-01 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Obesity
Keywords: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Part A: single-ascending dose Part B: multiple-ascending dose
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HM15275 (Experimental): Active comparator:
  Part A: single-ascending dose
  Single doses of HM15275 in healthy adults administered via subcutaneous injection.
  Part B: multiple-ascending dose
  Multiple doses of HM15275 in obese adults administered via subcutaneous injection.
  Interventions: Drug: HM15275; Drug: Placebo of HM15275
- Placebo of HM15275 (Placebo Comparator): Placebo comparator:
  Part A: single-ascending dose
  Single doses of HM15275 placebo in healthy adults administered via subcutaneous injection.
  Part B: multiple-ascending dose
  Multiple doses of HM15275 placebo in obese adults administered via subcutaneous injection.
  Interventions: Drug: HM15275; Drug: Placebo of HM15275

INTERVENTIONS:
Drug: HM15275 — HM15275 is a sterile solution for subcutaneous injection, supplied pre-filled syringes.
Drug: Placebo of HM15275 — A sterile, matching solution supplied in pre-filled syringes.

SUMMARY:
This Study is a Phase 1 Study to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of HM15275 in Healthy and Obese Subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Female and male adults, ages ≥ 18 and ≤ 65 years.
2. Part A: Healthy subjects with body mass index (BMI) ≥ 20.0 kg/m2 and ≤ 27 kg/m2.

   Part B: Obese subjects with BMI ≥ 30.0 kg/m2 and ≤ 45.0 kg/m2 with a stable body weight for 3 months prior to screening (defined as change < 5%).
3. HbA1c < 6.5 % [based on American Diabetes Association, 2023].
4. Female subjects must be non-pregnant and non-lactating.
5. Subjects must be able to provide written informed consent and are willing to follow study procedures and commitment to the study duration.

Exclusion Criteria:

1. Subject with existence of any surgical or medical condition that, in the judgment of the Investigator, might interfere with the absorption, distribution, metabolism or excretion of the investigational product.
2. Active or untreated malignancy or has been in remission from clinically significant malignancy (other than basal cell or squamous cell skin cancer, in situ carcinomas of the cervix, or in situ prostate cancer) for < 5 years.
3. Subjects with a history of any serious adverse reaction or hypersensitivity to study drug components (includes GLP-1, GIP, glucagon analogs) or have contraindicating diseases.
4. Subjects with confirmed type 1 or type 2 diabetes.
5. Subject is unwilling to avoid consumption of coffee and caffeine-containing beverages within from 24 hours before each study visit and while subjects are confined to the study center.
6. Subject is unwilling to abstain from vigorous exercise from 48 hours prior to admission until the Follow-up visit.
7. History of alcohol abuse as judged by the Investigator within approximately 1 year prior to Screening.
8. History of regular use (defined as ≥ 10 cigarettes per day) of nicotine-containing products (including but not limited to cigarettes, e-cigarettes, pipe, chewing tobacco, nicotine patch or gum) or vaping products within 6 weeks prior to check-in for the first In-house Period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2024-05-28 (Actual); Primary Completion 2025-05-02 (Actual); Study Completion 2025-05-02 (Actual)

PRIMARY OUTCOMES:
Part A: Safety and Tolerability | Up to Day 29
  Number of participants with treatment-emergent adverse events (TEAEs) after a single subcutaneous dose
Part B: Safety and Tolerability | Up to Day 57
  Number of participants with treatment-emergent adverse events (TEAEs) after multiple subcutaneous doses

SECONDARY OUTCOMES:
Part A: Pharmacokinetics | Up to Day 29
  Plasma concentration profile of HM15275 over time after a single subcutaneous dose
Part B: Pharmacokinetics | Up to Day 57
  Plasma concentration profile of HM15275 over time after multiple subcutaneous doses

OTHER OUTCOMES:
Part A: Pharmacodynamics | Up to Day 29
  Change in body weight (kg) from baseline
Part B: Pharmacodynamics | Up to Day 57
  Change in body weight (kg) from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- ProSciento, Inc., Chula Vista, California, United States

IPD SHARING:
Plan to Share IPD: Undecided